CLINICAL TRIAL: NCT03546907
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Proof-of-Concept (PoC) Study to Assess the Efficacy, Safety and Tolerability of SAR440340, in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Proof-of-Concept Study to Assess the Efficacy, Safety and Tolerability of SAR440340 (Anti-IL-33 mAb) in Patients With Moderate-to-severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACT15104; 2017-003290-34 (EudraCT Number); U1111-1194-2134 (Other: UTN)
Record Dates: First submitted 2018-05-17; First posted 2018-06-06 (Actual); Results first posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — itepekimab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo matched to SAR440340 administered as 2 subcutaneous (SC) injections every 2 weeks (Q2W). Participants were treated for a minimum of 24 weeks and up to a maximum of 52 weeks (last dose administered at Week 50, End of Treatment (EOT) visit occurred 2 weeks after last administration of IMP i.e., at Week 52).
  Interventions: Drug: Placebo; Drug: Any Inhaled Corticosteroids as prescribed by treating physician as standard of care; Drug: Any Long Acting Beta Agonist as prescribed by treating physician as standard of care; Drug: Any Long Acting Muscarinic Agonist as prescribed by treating physician as standard of care; Drug: Any short-acting β agonist as prescribed by treating physician as standard of care
- SAR440340 (Experimental): Participants received SAR440340 300 milligrams (mg) administered as 2 SC injections Q2W. Participants were treated for a minimum of 24 weeks and up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of IMP i.e., at Week 52).
  Interventions: Drug: SAR440340; Drug: Any Inhaled Corticosteroids as prescribed by treating physician as standard of care; Drug: Any Long Acting Beta Agonist as prescribed by treating physician as standard of care; Drug: Any Long Acting Muscarinic Agonist as prescribed by treating physician as standard of care; Drug: Any short-acting β agonist as prescribed by treating physician as standard of care

INTERVENTIONS:
Drug: SAR440340 — Pharmaceutical form: Solution for injection; Route of administration: SC
  Other Names: Itepekimab; REGN3500
  Arms: SAR440340
Drug: Placebo — Pharmaceutical form: Solution for injection; Route of administration: SC
  Arms: Placebo
Drug: Any Inhaled Corticosteroids as prescribed by treating physician as standard of care — Pharmaceutical form: Aerosol or Dry Powder inhaler Route of administration: Inhaled
Drug: Any Long Acting Beta Agonist as prescribed by treating physician as standard of care — Pharmaceutical form: Aerosol or Dry Powder inhaler; Route of administration: Inhaled
Drug: Any Long Acting Muscarinic Agonist as prescribed by treating physician as standard of care — Pharmaceutical form: Aerosol or Dry Powder inhaler; Route of administration: Inhaled
Drug: Any short-acting β agonist as prescribed by treating physician as standard of care — Pharmaceutical form: Aerosol or Dry Powder inhaler; Route of administration: inhaled

SUMMARY:
Primary Objective:

To investigate effects of SAR440340 (anti-interleukin-33 [IL-33] monoclonal antibody [mAb]) compared with placebo, on the annualized rate of moderate-to-severe acute exacerbations of COPD (AECOPD) over up to 52 weeks of treatment.

* Moderate exacerbations were recorded by the Investigator and defined as AECOPD that require either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics.
* Severe exacerbations were recorded by the Investigator and defined as AECOPD requiring hospitalization, emergency medical care visit or resulting in death.

Secondary Objectives:

To investigate effects of SAR440340 compared with placebo, on improving respiratory function, as assessed by pre-bronchodilator forced exploratory volume in 1 second (FEV1).

To evaluate effects of SAR440340 compared with placebo, on post-bronchodilator FEV1.

To evaluate effects of SAR440340 compared with placebo, on duration from baseline to first moderate or severe AECOPD event.

To evaluate effects of SAR440340 compared with placebo, on safety and tolerability.

DETAILED DESCRIPTION:
Study participation for each participant were up to a total of 46 weeks to 76 weeks including up to 10 days to 4 weeks of screening, 24-to-52 week treatment period on investigational medical product (IMP), and 20 weeks of post IMP treatment period.

ELIGIBILITY:
Inclusion criteria :

* Participants with a diagnosis of chronic obstructive pulmonary disease (COPD) for at least 1 year (based on Global Initiative for Chronic Obstructive Lung Disease [GOLD] definition).
* Participants with moderate-to-severe COPD (post-bronchodilator forced expiratory volume in 1 second [FEV1]/forced vital capacity [FVC] less than [<] 70 percent (%) and post-bronchodilator FEV1% predicted <80%, but greater than equal to [>=] 30%).
* Participants with COPD assessment test (CAT) score >=10 at Screening.
* Participants with reported history of signs and symptoms of chronic bronchitis (chronic productive cough for 3 months in the year up to screening in a participant in whom other causes of chronic cough [e.g., gastroesophageal reflux, chronic rhinosinusitis, bronchiectasis] had been excluded).
* Participants with a documented history (e.g., medical record verification) of >=2 moderate exacerbations or >=1 severe exacerbation within the year prior to screening. A moderate exacerbation was defined as an acute exacerbation of COPD (AECOPD) requiring systemic corticosteroids (oral, intravenous, or intramuscular) and/or treatment with antibiotics (however, use of antibiotics alone does not qualify as a "moderate exacerbation" unless documentation was available that use of antibiotics was necessary for treatment of worsening symptoms of COPD). A severe exacerbation was defined as an AECOPD that required a hospitalization.
* Participants with standard of care background therapy, for 3 months and at a stable dose for at least 1 month, including either:
* Double therapy: Long acting beta agonist (LABA) + Long acting muscarinic agonist (LAMA) or inhaled corticosteroid (ICS) + LABA or ICS + LAMA.

or

* Triple therapy: LABA + LAMA + ICS.
* Current or former smokers with a smoking history of >=10 packs/year.

Exclusion criteria:

* Concomitant severe diseases or diseases for which the use of ICS (e.g., active pulmonary tuberculosis, etc.) or LABA were contraindicated (e.g., diagnosis of a history of significant cardiovascular diseases, insulin-dependent diabetes mellitus, hyperthyroidism, thyrotoxicosis, pheochromocytoma, hypokalemia).
* Use of injectable glucocorticosteroids or oral systemic glucocorticosteroids within previous 1 month or more than 4 courses of intravenous glucocorticosteroids within the previous 6 months.
* Participants with bronchial thermoplasty procedure (up to 3 years prior to Visit 1).
* A current diagnosis of asthma according to the Global Initiative for Asthma (GINA) guidelines.
* Significant pulmonary disease other than COPD (e.g., lung fibrosis, sarcoidosis, interstitial lung disease, pulmonary hypertension, bronchiectasis, eosinophilic granulomatosis with polyangiitis, significant sleep apnea on Bilevel Positive Airway Pressure, etc.) or another diagnosed pulmonary or systemic disease associated with elevated peripheral eosinophil counts.
* Diagnosis of α-1 anti-trypsin deficiency.
* Advanced COPD with need for chronic (greater than [>] 15 hours/day) oxygen support.
* Participant with a moderate or severe acute exacerbation of COPD event within previous 4 weeks.
* A participant who has experienced an upper or lower respiratory tract infection within previous 4 weeks.
* Prior history of or planned pneumonectomy or lung volume reduction surgery.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2020-02-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (83):
- United States (16):
  - Investigational Site Number 8400002, Los Angeles, California
  - Investigational Site Number 8400003, Riverside, California
  - Investigational Site Number 8400006, Rolling Hills Estates, California
  - Investigational Site Number 8400015, Westminster, California
  - Investigational Site Number 8400013, Jacksonville, Florida
  - Investigational Site Number 8400012, Columbia, Maryland
  - Investigational Site Number 8400016, North Dartmouth, Massachusetts
  - Investigational Site Number 8400020, South Dartmouth, Massachusetts
  - Investigational Site Number 8400011, Minneapolis, Minnesota
  - Investigational Site Number 8400005, Jamaica, New York
  - Investigational Site Number 8400019, Chapel Hill, North Carolina
  - Investigational Site Number 8400004, Raleigh, North Carolina
  - Investigational Site Number 8400001, Medford, Oregon
  - Investigational Site Number 8400009, Philadelphia, Pennsylvania
  - Investigational Site Number 8400007, Plano, Texas
  - Investigational Site Number 8400008, Greenfield, Wisconsin
- Argentina (6):
  - Investigational Site Number 0320001, Buenos Aires
  - Investigational Site Number 0320005, Caba
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320004, Caba
  - Investigational Site Number 0320006, Quilmes
  - Investigational Site Number 0320003, Rosario
- Australia (6):
  - Investigational Site Number 0360005, Bedford Park
  - Investigational Site Number 0360002, Chermside
  - Investigational Site Number 0360004, Clayton
  - Investigational Site Number 0360003, Frankston
  - Investigational Site Number 0360006, Kent Town
  - Investigational Site Number 0360001, Murdoch
- Canada (9):
  - Investigational Site Number 1240002, Burlington
  - Investigational Site Number 1240009, Hamilton
  - Investigational Site Number 1240003, Montreal
  - Investigational Site Number 1240001, Montreal
  - Investigational Site Number 1240005, Québec
  - Investigational Site Number 1240006, Saint-Charles-Borromée
  - Investigational Site Number 1240008, Trois-Rivières
  - Investigational Site Number 1240007, Vancouver
  - Investigational Site Number 1240004, Victoriaville
- Chile (6):
  - Investigational Site Number 1520002, Quillota
  - Investigational Site Number 1520001, Santiago
  - Investigational Site Number 1520007, Santiago
  - Investigational Site Number 1520004, Santiago
  - Investigational Site Number 1520005, Talca
  - Investigational Site Number 1520003, Talcahuano
- Germany (6):
  - Investigational Site Number 2760006, Berlin
  - Investigational Site Number 2760001, Großhansdorf
  - Investigational Site Number 2760002, Hamburg
  - Investigational Site Number 2760007, Koblenz
  - Investigational Site Number 2760004, München
  - Investigational Site Number 2760005, Rüdersdorf Bei Berlin
- Poland (9):
  - Investigational Site Number 6160001, Bialystok
  - Investigational Site Number 6160008, Bialystok
  - Investigational Site Number 6160005, Bydgoszcz
  - Investigational Site Number 6160009, Grudziądz
  - Investigational Site Number 6160007, Krakow
  - Investigational Site Number 6160002, Poznan
  - Investigational Site Number 6160006, Poznan
  - Investigational Site Number 6160010, Rzeszów
  - Investigational Site Number 6160003, Żnin
- Russia (9):
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430005, Moscow
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430007, Saint Petersburg
  - Investigational Site Number 6430010, Saint Petersburg
  - Investigational Site Number 6430006, Saint Petersburg
  - Investigational Site Number 6430009, Stavropol
  - Investigational Site Number 6430004, Ulyanovsk
- Turkey (Türkiye) (6):
  - Investigational Site Number 7920004, Ankara
  - Investigational Site Number 7920001, Istanbul
  - Investigational Site Number 7920006, Izmir
  - Investigational Site Number 7920007, Izmir
  - Investigational Site Number 7920008, Kırıkkale
  - Investigational Site Number 7920002, Mersin
- Ukraine (10):
  - Investigational Site Number 8040008, Chernivtsi
  - Investigational Site Number 8040012, Ivano-Frankivsk
  - Investigational Site Number 8040004, Ivano-Frankivsk
  - Investigational Site Number 8040002, Kharkiv
  - Investigational Site Number 8040011, Kharkiv
  - Investigational Site Number 8040007, Kyiv
  - Investigational Site Number 8040001, Kyiv
  - Investigational Site Number 8040006, Odesa
  - Investigational Site Number 8040003, Ternopil
  - Investigational Site Number 8040005, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Rabe KF, Celli BR, Wechsler ME, Abdulai RM, Luo X, Boomsma MM, Staudinger H, Horowitz JE, Baras A, Ferreira MA, Ruddy MK, Nivens MC, Amin N, Weinreich DM, Yancopoulos GD, Goulaouic H. Safety and efficacy of itepekimab in patients with moderate-to-severe COPD: a genetic association study and randomised, double-blind, phase 2a trial. Lancet Respir Med. 2021 Nov;9(11):1288-1298. doi: 10.1016/S2213-2600(21)00167-3. Epub 2021 Jul 21. PMID 34302758

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 83 centers in 10 countries, out of which 78 centers randomized at least 1 participant. A total of 653 participants were screened from 16-July-2018 to 01-April-2019, of which 310 participants were screen failures mainly due to selection criteria not met.
Pre-assignment Details: A total of 343 participants were randomized and treated in this study. Participants were randomized in 1:1 ratio to receive treatment SAR440340 and matching placebo for SAR440340.
Groups:
- Placebo: Participants received placebo matched to SAR440340 administered as 2 subcutaneous (SC) injections every 2 weeks (Q2W). Participants were treated for a minimum of 24 weeks and up to a maximum of 52 weeks (last dose administered at Week 50, End of Treatment [EOT] visit occurred 2 weeks after last administration of investigational medicinal product [IMP] i.e., at Week 52).
Period: Overall Study
Arm/Group | Placebo | SAR440340
Started | 171 | 172
Completed | 154 | 151
Not Completed | 17 | 21
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 8 | 9
Not completed — Adverse events (AEs) | 7 | 10
Not completed — Other-unspecified | 1 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population included any participant who had signed informed consent and had been allocated to a randomized treatment regardless of whether the treatment kit was used.
Groups:
- Placebo: Participants received placebo matched to SAR440340 administered as 2 SC injections Q2W. Participants were treated for a minimum of 24 weeks and up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of IMP i.e., at Week 52).
- SAR440340: Participants received SAR440340 300 mg administered as 2 SC injections Q2W. Participants were treated for a minimum of 24 weeks and up to a maximum of 52 weeks (last dose administered at Week 50, EOT visit occurred 2 weeks after last administration of IMP i.e., at Week 52).
- Total: Total of all reporting groups
Arm/Group | Placebo | SAR440340 | Total
Number analyzed (Participants) | 171 | 172 | 343
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (6.5) | 63.7 (6.8) | 63.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 76 | 73 | 149
  Male | 95 | 99 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 169 | 170 | 339
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Age at diagnosis of chronic obstructive pulmonary disease (COPD) [Mean (Standard Deviation); unit: years] | 55.5 (8.0) | 55.4 (7.8) | 55.4 (7.9)
Mean number of moderate COPD exacerbations experienced within 1 year before screening visit [Mean (Standard Deviation); unit: exacerbations] — Moderate exacerbations events were defined as acute exacerbation of chronic obstructive pulmonary disease (AECOPD) that require either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics.
  exacerbations | 1.8 (1.2) | 1.8 (1.1) | 1.8 (1.2)
Mean number of severe COPD exacerbations experienced within 1 year before screening visit [Mean (Standard Deviation); unit: exacerbations] — Severe exacerbations events were defined as AECOPD requiring hospitalization, emergency medical care visit or resulting in death.
  exacerbations | 0.4 (0.6) | 0.3 (0.6) | 0.4 (0.6)
Number of participants with smoking history [Count of Participants; unit: Participants] — Participants with current and former smoking history status were reported in this baseline measure.
  Participants
    Current | 82 | 74 | 156
    Former | 89 | 98 | 187
Predicted baseline post-bronchodilator (BD) forced expiratory volume in 1 second (FEV1) [Mean (Standard Deviation); unit: percent predicted FEVI] — FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer.
  percent predicted FEVI | 49.02 (12.18) | 49.62 (12.34) | 49.32 (12.25)
Baseline COPD assessment test (CAT) score [Mean (Standard Deviation); unit: score on a scale] — The CAT is a 8-item self-administered questionnaire that is designed for participants with COPD to measure the effects of the disease on their quality of lives. Each question is scored in a range between 0 to 5 according to participant feelings about the disease, where 0 = "I am very happy" to 5 = "I am very sad". Total CAT score (sum of the 8 individual question scores) ranged from 0 to 40, where 0 to 10= mild, 11 to 20= moderate, 21 to 30= severe, 31 to 40= very severe; higher score indicated worse symptoms.
  score on a scale | 21.66 (5.23) | 21.89 (5.84) | 21.78 (5.54)
Standard of care background therapy [Count of Participants; unit: Participants] — At screening, participants were on standard of care background therapy, for 3 months prior to Visit 2/Randomization and at a stable dose for at least 1 month prior to the Screening Visit 1, including either: Double therapy: long-acting beta2 [β2] adrenergic agonist (LABA) + Long-acting muscarinic antagonist (LAMA) or inhaled corticosteroid (ICS) + LABA or ICS + LAMA; or Triple therapy: ICS + LABA + LAMA.
  Participants
    LABA+LAMA | 26 | 23 | 49
    ICS+LABA | 34 | 33 | 67
    ICS+LAMA | 0 | 1 | 1
    ICS+LABA+LAMA | 111 | 115 | 226
Baseline blood eosinophil count [Mean (Standard Deviation); unit: Giga cells per liter] | 0.25 (0.19) | 0.27 (0.24) | 0.26 (0.22)

OUTCOME MEASURES:

1. Primary Outcome: Annualized Rate of Moderate to Severe Acute Exacerbation Events in Chronic Obstructive Pulmonary Disease (AECOPD) Participants
Description: Moderate exacerbations events were recorded by the investigator and defined as AECOPD that require either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations events were defined as AECOPD requiring hospitalization, emergency medical care visit or resulting in death. Annualized event rate was the total number of exacerbations that occurred during the treatment period divided by the total number of participant-years treated.
Time Frame: From Baseline up to Week 52
Population: Analysis was performed on modified intent-to-treat (mITT) population that included all randomized participants who had received at least 1 dose of IMP, analyzed according to the treatment group allocated by randomization.
Measure: Number (95% Confidence Interval); unit: exacerbation per participant-year
Arm/Group | Placebo | SAR440340
Number analyzed (Participants) | 171 | 172
exacerbation per participant-year | 1.610 [1.318 to 1.968] | 1.301 [1.052 to 1.61]
Statistical Analysis 1: Comparison: Placebo vs SAR440340; Analysis was performed using negative binomial regression model with total number of events occurring during observation duration as response variable, treatment, baseline eosinophil strata, region, number of severe COPD exacerbations experienced in previous year(0 vs. 1+) at baseline, smoking history(current vs. former smoker), post-BD FEV1 percent(%) predicted (less than[<] 50% vs greater than equal[>=]50%) at baseline as covariates, and log-transformed observation duration as offset variable; Test type: Superiority; p = 0.1296, Negative binomial regression model; Risk Ratio (RR) = 0.808, 95% CI 2-sided [0.613 to 1.065]

2. Secondary Outcome: Average Change in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) From Baseline to Week 16 Through Week 24
Description: FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Spirometry was performed after a wash out period of bronchodilators according to their action duration. A mixed-effect model with repeated measures (MMRM) was first used to model the change from baseline at each post randomization timepoint up to Week 24, then the predicted values of Week 16 to Week 24 were averaged to provide an overall assessment of change from baseline in FEV1.
Time Frame: From Baseline to Week 16 through Week 24
Population: Analysis was performed on mITT population.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | SAR440340
Number analyzed (Participants) | 171 | 172
liters | 0.0 (0.02) | 0.06 (0.02)

3. Secondary Outcome: Change From Baseline in Post-bronchodilator Forced Expiratory Volume (FEV1) in 1 Second at Week 24
Description: FEV1 was the volume of air exhaled from the lungs in the first second of a forced expiration as measured by spirometer. Post-bronchodilator FEV1 referred to the spirometry performed within 30 minutes after administration of bronchodilator (4 puffs of salbutamol/albuterol [100 micrograms {mcg}] or ipratropium bromide [20 mcg]).
Time Frame: Baseline, Week 24
Population: Analysis was performed on mITT population. Here, 'Overall number of participants analyzed ' signifies number of participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | SAR440340
Number analyzed (Participants) | 163 | 165
liters | 0.01 (0.22) | 0.04 (0.24)

4. Secondary Outcome: Time to First Moderate or Severe Acute Exacerbation of Chronic Obstructive Pulmonary Disease (AECOPD)
Description: The time to first moderate or severe exacerbation was defined as onset date of first moderate or severe AECOPD minus randomization date + 1. The median time to first severe exacerbation was derived from Kaplan-Meier estimates. Moderate exacerbations events were recorded by the investigator and defined as AECOPD that require either systemic corticosteroids (such as intramuscular, intravenous or oral) and/or antibiotics. Severe exacerbations events were defined as AECOPD requiring hospitalization, emergency medical care visit or resulting in death.
Time Frame: From Baseline up to 52 weeks
Population: Analysis was performed on mITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | SAR440340
Number analyzed (Participants) | 171 | 172
days | 199.0 [139.00 to 266.00] | 277.0 [204.00 to NA] — Here, 'NA' signifies that the upper limit of 95% confidence interval was not computable because the curve that represents the upper confidence limits for the survivor function lies above 0.5.

ADVERSE EVENTS:
Time Frame: From first administration of IMP up to 22 weeks after last dose of IMP (i.e., minimum up to 46 weeks and a maximum of up to 72 weeks) regardless of seriousness or relationship to IMP
Description: Analysis was performed on safety population that included all randomized participants who received at least 1 injection of IMP.
Arm/Group | Placebo | SAR440340
All-Cause Mortality (participants affected / at risk) | 2/171 | 3/172
Serious Adverse Events (participants affected / at risk) | 36/171 | 29/172
Other Adverse Events (participants affected / at risk) | 78/171 | 60/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=171) | SAR440340 (N=172)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 1 (1) | 2 (2)
Cardio-Respiratory Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary Failure (Cardiac disorders) | 0 (0) | 1 (1)
Coronary Artery Stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 1 (2) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1)
Chronic Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Obstructive Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis Chronic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0)
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Babesiosis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Cellulitis Of Male External Genital Organ (Infections and infestations) | 0 (0) | 1 (1)
Cholecystitis Infective (Infections and infestations) | 0 (0) | 1 (1)
Infective Exacerbation Of Chronic Obstructive Airways Disease (Infections and infestations) | 5 (7) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3) | 2 (2)
Pneumonia Pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pulmonary Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (2) | 0 (0)
Subperiosteal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Burns Second Degree (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Facial Paresis (Nervous system disorders) | 0 (0) | 1 (1)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 1 (1)
Thrombotic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 2 (2) | 0 (0)
Alcohol Abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (1)
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 14 (19) | 11 (12)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pickwickian Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=171) | SAR440340 (N=172)
Bronchitis (Infections and infestations) | 14 (17) | 16 (20)
Nasopharyngitis (Infections and infestations) | 29 (43) | 28 (40)
Upper Respiratory Tract Infection (Infections and infestations) | 14 (17) | 13 (17)
Headache (Nervous system disorders) | 23 (35) | 14 (24)
Hypertension (Vascular disorders) | 11 (12) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/07/NCT03546907/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT03546907/SAP_001.pdf